CLINICAL TRIAL: NCT04415671
Title: A Phase 1, Dose-escalating Study of the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Doses of AD-214 When Administered Intravenously to Healthy Volunteers
Brief Title: Phase 1 Safety, Tolerability, PK & PD Study of AD-214 Administered to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AdAlta Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADA-AD-214-1A
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: SAD Part A in HVs- Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) MAD Part B in HVs- Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A- AD-214 SAD in Healthy Volunteers (Experimental)
  Interventions: Biological: AD-214
- Part A-Placebo SAD in Healthy Volunteers (Placebo Comparator)
  Interventions: Other: Placebo
- Part B-AD-214 MAD in Healthy Volunteers (Experimental)
  Interventions: Biological: AD-214
- Part B-Placebo MAD in Healthy Volunteers (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AD-214 — AD-214 is a recombinant Fc-fusion protein that selectively binds to CXCR4 to antagonise the SDF-1/CXCR4 axis.
  Arms: Part A- AD-214 SAD in Healthy Volunteers; Part B-AD-214 MAD in Healthy Volunteers
Other: Placebo — Placebo
  Arms: Part A-Placebo SAD in Healthy Volunteers; Part B-Placebo MAD in Healthy Volunteers

SUMMARY:
This is a first in human (FIH), multi-center, dose escalating study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of AD-214 when administered to healthy volunteers (HVs). The study in HVs will be a randomized, double blind, and placebo-controlled single ascending dose (SAD) and multiple ascending dose (MAD) (Part B) study.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide signed informed consent prior to study entry and agree to adhere to all study protocol requirements.
2. Maximum weight of 100 kg at the time of consent and body mass index (BMI) >18 and < 30 kg/m2 (inclusive)
3. Must agree to abstain from alcohol intake from 48 hours before first study drug administration through to final study visit
4. Must agree to abstain from smoking from 48 hours before first study drug administration through to final study visit
5. Must have a negative urine drug screen and cotinine test, and alcohol breath test at Screening and on Day -1 (admission).
6. Must agree to use highly effective, double barrier contraception (both male and female partners) at least 30 days prior to dosing on day 1, during the study AND for 90 days following completion of dosing
7. Male participants must refrain from sperm donation from start of study and for 90 days after last dose of AD-214
8. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.
9. Participants must be in good general health, with no significant medical history, and no clinically significant abnormalities on physical examination at Screening, and/or before administration of the initial dose of study drug.
10. Participants must have clinical laboratory values within normal range or < 1.5 x upper limit of normal (ULN) as specified by the testing laboratory at Screening.

Exclusion Criteria:

1. Received any Investigational Medicinal Product (IMP) within 30 days (4 months if the previous drug was a new chemical entity) or 5 half-lives prior to Screening
2. Received an investigational vaccine within 6 months, a live attenuated vaccine within 60 days or a registered vaccine within 30 days prior to the first dose of the investigational product.
3. Received blood products within 1 month prior to Screening.
4. Blood donation or significant blood loss (> 450 mL) within 60 days prior to the first administration of investigational product
5. Plasma donation within 7 days prior to the first administration of investigational product.
6. A bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with blood draws.
7. Known history of Human Immunodeficiency Virus (HIV) or HIV antibody positive.
8. Hepatitis B surface Antigen (HBsAg) positive or Hepatitis B Virus (HBV) polymerase chain reaction (PCR) positivity. Hepatitis C Virus (HCV) antibody positive or HCV PCR positivity.
9. Any clinically significant abnormality at Screening determined by medical history, physical examination, blood chemistry, hematology, coagulation, urinalysis and 12-lead electrocardiogram (ECG).
10. A history of or current clinically significant gastrointestinal, hepatic, renal, cardiovascular, respiratory (apart from ILD), endocrine, oncological, immunodeficiency, neurological, metabolic, hematological, autoimmune or social or psychiatric condition which in the investigator's opinion may interfere with the study objectives, may put the participant at risk or may make the participant unsuitable for participation in the study.
11. Surgery within the past 3 months prior to the first study drug administration determined by the PI to be clinically relevant.
12. History or presence of alcohol or drug abuse
13. Females who are pregnant or lactating.
14. Use of any prescription or over the counter medication (with the exception of paracetamol and contraceptives) within 7 days of first study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as assessed by the number of abnormal laboratory values and/or adverse events that are related to treatment | SAD Part A- 28 days. MAD Part B - 57 days

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - CMAX Clinical Research Pty Ltd, Adelaide, South Australia